CLINICAL TRIAL: NCT01055977
Title: Statin Therapy Results in the Real World Practice in the Czech Republic
Acronym: STEP
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CCZ-CRE-2009/1
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Dyslipidaemia
Keywords: statin therapy; treatment goal; dyslipidaemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Statins are the first choice treatment of dyslipidemia, a major contributor to cardiovascular diseases. Statins also have enough evidence to demonstrate decrease of morbidity and mortality from cardiovascular diseases. Even though statin therapy is effective treatment of dyslipidaemia not all patients reach the goal levels.

The aim of the study is to estimate proportion of patients who achieved the therapeutic goal (LDL-C. total cholesterol, HDL-C and triglycerides levels) after at least one year of a statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Documented statin therapy for at least 12 months
* Available two LDL-C values: one at the beginning of statin therapy or at the time when patient comes to a specialist; and the other one at least after 12 months of treatment. The latter value should not be older than 6 months.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: specialist care clinics
Sampling Method: Probability Sample
Enrollment: 3253 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
LDL-C | one year

SECONDARY OUTCOMES:
Total cholesterol | one year
HDL-C | one year
triglycerides | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ales Kminek, Study Director — AstraZeneca; Jaromir Hradec, Principal Investigator — General faculty hospital Prague; Jan Bultas, Principal Investigator — Faculty hospital Kralovske Vinohrady Prague
Locations (95):
- Czechia (95):
  - Research Site, Benešov
  - Research Site, Beroun
  - Research Site, Blansko
  - Research Site, Bohumín
  - Research Site, Boskovice
  - Research Site, Brandýs nad Labem
  - Research Site, Brno
  - Research Site, Cheb
  - Research Site, Chomutov
  - Research Site, Chrudim
  - Research Site, Česká Lípa
  - Research Site, České Budějovice
  - Research Site, Český Krumlov
  - Research Site, Děčín
  - Research Site, Domažlice
  - Research Site, Dvůr Králové nad Labem
  - Research Site, Fryštát
  - Research Site, Frýdek-Místek
  - Research Site, Havířov
  - Research Site, Havlíčkův Brod
  - Research Site, Hradec Králové
  - Research Site, Hustopeče
  - Research Site, Ivančice
  - Research Site, Jablonec nad Nisou
  - Research Site, Jeseník
  - Research Site, Jičín
  - Research Site, Jihlava
  - Research Site, Jindřichův Hradec
  - Research Site, Karlovy Vary
  - Research Site, Kladno
  - Research Site, Kolín
  - Research Site, Krnov
  - Research Site, Kuřim
  - Research Site, Kutná Hora
  - Research Site, Kyjov
  - Research Site, Liberec
  - Research Site, Litoměřice
  - Research Site, Louny
  - Research Site, Mělník
  - Research Site, Městec Králové
  - Research Site, Mikulov
  - Research Site, Milevsko
  - Research Site, Mladá Boleslav
  - Research Site, Moravská Třebová
  - Research Site, Moravské Budějovice
  - Research Site, Moravský Krumlov
  - Research Site, Most
  - Research Site, Náchod
  - Research Site, Nový Bydžov
  - Research Site, Olomouc
  - Research Site, Opava
  - Research Site, Orlová
  - Research Site, Ostrava
  - Research Site, Ostrov
  - Research Site, Pardubice
  - Research Site, Pelhřimov
  - Research Site, Pilsen
  - Research Site, Písek
  - Research Site, Police nad Metují
  - Research Site, Polička
  - Research Site, Prachatice
  - Research Site, Prague
  - Research Site, Prostějov
  - Research Site, Přerov
  - Research Site, Přeštice
  - Research Site, Příbram
  - Research Site, Rakovník
  - Research Site, Roudnice nad Labem
  - Research Site, Rožnov pod Radhoštěm
  - Research Site, Rychnov nad Kněžnou
  - Research Site, Semily
  - Research Site, Slaný
  - Research Site, Smiřice
  - Research Site, Sternberk
  - Research Site, Strakonice
  - Research Site, Sušice
  - Research Site, Svitavy
  - Research Site, Tábor
  - Research Site, Teplice
  - Research Site, Tišnov
  - Research Site, Trutnov
  - Research Site, Třebíč
  - Research Site, Třinec
  - Research Site, Turnov
  - Research Site, Uherské Hradiště
  - Research Site, Ústí nad Labem
  - Research Site, Valašské Klobouky
  - Research Site, Veselí nad Moravou
  - Research Site, Vítkovice
  - Research Site, Vsetín
  - Research Site, Vysoké Mýto
  - Research Site, Vyškov
  - Research Site, Zlín
  - Research Site, Znojmo
  - Research Site, Žamberk